CLINICAL TRIAL: NCT07385144
Title: A Pilot Study Evaluating the Effects of a Dietary Supplement on Serum Biomarkers in Children
Brief Title: A Study of a Dietary Supplement on Serum Biomarkers in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SF Research Institute, Inc. (Network)
Collaborators: Smarty Pants Vitamins (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPV20251119 - 01
Record Dates: First submitted 2026-01-27; First posted 2026-02-03 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Nutritional Status; Serum Biomarkers
Keywords: Dietary Supplement; Pediatric Nutrition; Nutritional Biomarkers; Vitamins; Omega-3 Fatty Acids; Vitamin D; Vitamin B12
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary Supplement Group (Experimental): Participants in this arm will receive the investigational dietary supplement (Kids Multi & Omegas) in gummy form. Subjects will be instructed to take two gummies once daily, with or without food, for a total duration of 4 weeks. Blood samples will be collected at baseline and at the end of the study to evaluate changes in selected serum nutritional biomarkers.
  Interventions: Dietary Supplement: Dietary Supplement (Kids Multi & Omegas)

INTERVENTIONS:
Dietary Supplement: Dietary Supplement (Kids Multi & Omegas) — The intervention consists of a gummy dietary supplement administered orally to healthy children. Participants will be instructed to take two gummies once daily, with or without food, starting on Day 1 and continuing for a total duration of 4 weeks. The supplement contains vitamins, minerals, and omega-3 fatty acids, including vitamin D, vitamin B12, folate, and polyunsaturated fatty acids (DHA and EPA). The intervention is evaluated by measuring serum nutritional biomarkers at baseline and after 4 weeks of supplementation.
  Other Names: SPV20251119 - 01; Product A

SUMMARY:
This is a pilot clinical study designed to evaluate the effects of a dietary supplement on selected blood-based nutritional biomarkers in healthy children aged 4 to 15 years.

Approximately 24 children will be screened and enrolled to account for potential dropouts, with a target of 20 participants completing the study. Eligible participants will attend a screening and baseline visit, followed by daily intake of the study supplement for 4 weeks. After the supplementation period, participants will return to the clinic for an end-of-study visit.

Blood samples will be collected at baseline and after 4 weeks to measure nutritional biomarkers, including vitamin D, vitamin B12, folate, omega-3 fatty acids, and standard blood count parameters. Additional assessments include height, weight, body mass index (BMI), and a socioeconomic questionnaire. Throughout the study, participants or their caregivers will record daily supplement intake, any medications taken, and any adverse events in a study diary.

The results of this pilot study will provide preliminary data on the effects of the dietary supplement on serum biomarkers in children.

DETAILED DESCRIPTION:
This is a prospective, monadic pilot clinical study designed to evaluate the effects of a dietary supplement on serum nutritional biomarkers in healthy children. The study will be conducted at a single site, SF Research Institute, San Francisco, California.

Approximately 24 participants will be recruited to compensate for potential dropouts, with a target of 20 participants completing the study. Children aged 4 to 15 years who meet all inclusion and exclusion criteria will be eligible to participate. Recruitment will occur through the SF Research Institute database, social media, and public flyers.

The study consists of two clinic visits over a total study duration of approximately 4 weeks. At the Screening/Baseline Visit (Day 1), written informed consent from the parent or legal guardian and assent from the child will be obtained prior to any study procedures. Demographic information, medical history, socioeconomic status, and medication use will be collected, and eligibility criteria will be reviewed. Baseline anthropometric measurements, including height, weight, and body mass index (BMI), will be recorded.

At the baseline visit, participants will undergo phlebotomy for the collection of blood samples to assess nutritional biomarkers. Following completion of baseline assessments, eligible participants will be enrolled and provided with the investigational dietary supplement along with instructions for daily use over a 4-week period. Participants will also receive a daily diary to record supplement intake, concomitant medications (if taken), treatment compliance, and any adverse events.

The investigational product is a gummy dietary supplement, and participants will be instructed to take two gummies once daily, with or without food, starting on Day 1 and continuing for the duration of the study.

At the End-of-Study Visit (Week 4), participants will return to the clinic for review of the completed daily diary and assessment of compliance. A second blood sample will be collected for post-intervention biomarker analysis. Following completion of these procedures, participants will be discharged from the study.

Biomarker analyses will include measurements of 25-hydroxyvitamin D, serum vitamin B12, red blood cell folate, polyunsaturated fatty acids (including DHA and EPA), and a complete blood count. All laboratory analyses will be performed at Empire City Laboratories, Brooklyn, New York, USA.

All participants and their parents or guardians will have the opportunity to review the results of bloodwork, and instructions will be provided on how to contact the study physician for result-related questions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male and Females aged 4 - 15 years
* NORMAL BMI /growth (per CDC growth tables) Between 5th - 85th percentile.
* Able to read, understand, and complete the study questionnaire and records.
* Able to understand the study procedures.
* Able to comply with all study requirements.
* Written informed consent/Assent to participate in the study.
* Agrees to maintain current lifestyle habits (diet, physical activity, medications, and sleep) as much as possible throughout the study and avoid taking new supplements
* Willingness to actively participate in the study and to come to the scheduled visits.

Exclusion Criteria:

* Immune insufficiency
* Use of systemic corticosteroids or immunosuppressant drugs.
* Any diseases or medications that might directly interfere in the study or put the subject's health under risk.
* Currently taking any prescription medications or any dietary supplements including multivitamins
* Employees of the institute or the brand owner or the manufacturers of the product
* Cardiovascular-, chronic liver-, thyroid or kidney diseases; a history of cancer; a disease or condition that could influence the participants' ability to follow the study protocol,

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-05 (Estimated)

PRIMARY OUTCOMES:
Change in Serum 25-Hydroxyvitamin D From Baseline to Week 4 | Baseline (Day 1) and End of Study (Week 4)
  Change from baseline to Week 4 in serum 25-hydroxyvitamin D (25[OH]D), measured by phlebotomy as a marker of vitamin D status.
Change in Serum Vitamin B12 From Baseline to Week 4 | Baseline (Day 1) and End of Study (Week 4)
  Change from baseline to Week 4 in serum vitamin B12 (cobalamin) levels, measured by blood sample collection.
Change in Red Blood Cell Folate From Baseline to Week 4 | Baseline (Day 1) and End of Study (Week 4)
  Change from baseline to Week 4 in red blood cell (RBC) folate levels, measured by phlebotomy.
Change in Plasma Omega-3 Fatty Acids From Baseline to Week 4 | Baseline (Day 1) and End of Study (Week 4)
  Change from baseline to Week 4 in plasma polyunsaturated fatty acids, including docosahexaenoic acid (DHA) and eicosapentaenoic acid (EPA), measured by blood sample collection.
Change in Complete Blood Count Parameters From Baseline to Week 4 | Baseline (Day 1) and End of Study (Week 4)
  Change from baseline to Week 4 in complete blood count (CBC) parameters, including red blood cell count, hemoglobin, hematocrit, white blood cell count, and platelet count.

SECONDARY OUTCOMES:
Change in Body Mass Index From Baseline to Week 4 | Baseline (Day 1) and End of Study (Week 4)
  Change from baseline to Week 4 in body mass index (BMI), calculated using measured height and weight and compared with CDC growth tables for children.
Change in Height and Weight From Baseline to Week 4 | Baseline (Day 1) and End of Study (Week 4)
  Change from baseline to Week 4 in anthropometric measurements, including height and body weight, measured using a calibrated digital medical scale.
Socioeconomic Status Assessment at Baseline | Baseline (Day 1)
  Assessment of socioeconomic status using a structured questionnaire evaluating household income, parental education, living conditions, and access to resources.
Treatment Compliance and Diary Completion Over 4 Weeks | Baseline (Day 1) through End of Study (Week 4)
  Assessment of treatment compliance based on daily diary entries documenting supplement intake, concomitant medications (if taken), and study product use over the 4-week study period.
Incidence of Adverse Events During the Study Period | Baseline (Day 1) through End of Study (Week 4)
  Monitoring and documentation of adverse events reported by participants or caregivers during the 4-week supplementation period.

CONTACTS AND LOCATIONS:
Locations (1):
- San Francisco Research Institute, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No